CLINICAL TRIAL: NCT06472570
Title: Escalating a Biological Dose of Radiation in the Target Volume Applying Stereotactic Radiosurgery in Patients With Head and Neck Region Tumours
Brief Title: Stereotactic Radiosurgery in Patients With Head and Neck Region Tumours
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SterRad
Record Dates: First submitted 2024-05-21; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-05

CONDITIONS: Head and Neck Cancer
Keywords: stereotactic radiotherapy; radiosurgery boost; head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic radiotherapy (Experimental): Patients treated with stereotactic radiosurgery boost. Treatment is conducted as radiotherapy alone or radiochemotherapy based on cisplatin
  Interventions: Radiation: Stereotactic radiotherapy boost

INTERVENTIONS:
Radiation: Stereotactic radiotherapy boost — A stereotactic radiosurgery boost is given in two cases:
  * Upfront boost-on the first day of overall treatment time (OTT) (to 6 days before beginning conventional radiotherapy).
  * Direct boost-on Days 43-49 of OTT in relation to conventional radiotherapy to total dose (TD) 70 Gy, i.e., up to 6 days after a dose of 60 Gy.
  Treatment is conducted as radiotherapy alone or radiochemotherapy based on cisplatin 100 mg/m2 or 40 mg/m2 in a 21-day or 7-day cycle, respectively
  Patients who start the treatment from induction chemotherapy may have a chance to qualify for an upfront or direct boost, depending the evaluation of the response to systemic treatment
  Prescribed doses of stereotactic boost are in the range of 10-18 Gy

SUMMARY:
The goal of this study is to evaluate the safety and efficacy of the stereotactic boost applied in patients with H&N tumours.

DETAILED DESCRIPTION:
Aims of the study:

1. Evaluation of the efficacy of the stereotactic boost applied in patients with head and neck tumours.
2. Evaluation of the safety of the stereotactic boost applied in patients with head and neck tumours.
3. Evaluation of the influence of the stereotactic radiotherapy boost on blood parameters reflecting tumour response (interleukin 6 (Il-6), thymidine kinase (TK), Fms-related tyrosine kinase 1 (sFlt-1)), and normal tissue response (C-reactive protein (CRP)).

In the case of beneficial findings, the stereotactic radiosurgery boost in the course of radio(chemo)therapy in patients with head and neck tumours will be able to replace traditional techniques of radiation, and radical schemes of treatment will be possible for future development.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with squamous cell carcinoma (SCC) or adenoid cystic carcinoma (ACC) of the H&N region qualified for radical treatment with (definitive or adjuvant (adjuvant radiotherapy or radiochemotherapy in postoperative cases of R2 resection or early locoregional recurrence unsuitable for reoperation)) radiotherapy or radiochemotherapy.
2. Patients with other malignant tumours of the H&N region (sarcomas, neuroendocrine carcinomas, differentiated carcinomas, undifferentiated carcinomas, or basaloid carcinomas) qualified for radical treatment with (definitive or adjuvant (adjuvant radiotherapy or radiochemotherapy in postoperative cases of R2 resection or early locoregional recurrence unsuitable for reoperation)) radiotherapy or radiochemotherapy.
3. Patients with nonmalignant tumours of the H&N region (tumour mixtus or paraganglioma) demanding definitive or adjuvant radiotherapy.
4. Age: 18-80 years. Biomedicines 2022, 10, 1484 5 of 12
5. Performance status: Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
6. Conscious agreement to participate in the clinical trial.

Exclusion Criteria:

1. Do not meet the inclusion criteria.
2. Decompensated diabetes mellitus.
3. Myocardial infarction occurred up to 6 months before.
4. Pregnancy.
5. Mental disorder preclusive of making a conscious agreement

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-10-26 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Response to treatment | one month after the end of treatment, every 3 months in the first year, every 4 months in the second year, and every six months in the third-fifth years
  Response to treatment in imaging tests and clinical examination-local control (LC) and locoregional control (LRC).

SECONDARY OUTCOMES:
Evaluation of efficacy | 5 years after the end of treatment
  Evaluation of overall survival (OS) time
Evaluation of efficacy | 5 years after the end of treatment
  Evaluation of progression-free survival time (PFS)
Evaluation of efficacy | 5 years after the end of treatment
  Evaluation of disease-free survival time (DFS)
Evaluation of safety Terminology Criteria for Adverse Events (CTCAE)v4.0. | 5 years after the end of treatment
  Acute and late side effects according to the Common Terminology Criteria for Adverse Events (CTCAE) v 4.0.
Treatment tolerance | an average of 3 months
  Evaluation of quality of live anf reatment tolerance using QLQ-C30 (Quality of Life Questionnaire C30).

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Polanowski, Principal Investigator — Maria Sklodowska-Curie National Research Institute of Oncology in Gliwice
Locations (1):
- 1st Radiation and Clinical Oncology Department, Maria Sklodowska-Curie National Research Institute of Oncology, Gliwice Branch,, Gliwice, Gliwicw, Poland